CLINICAL TRIAL: NCT07383220
Title: Effect of Combined Transcutaneous Electrical Stimulation and Isometric Exercise on Peripheral Hemodynamic Parameters in Patients With Resistant Hypertension
Brief Title: Effect of Electrical Stimulation and Exercise on Blood Flow in Patients With Resistant High Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohamed Mohamed Ali Morgan (Other)
Responsible Party: Sponsor-Investigator, Mohamed Mohamed Ali Morgan, Demonstrator of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006060
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Resistant Hypertension; Hemodynamic Instability; Essential (Primary) Hypertension; Abdominal Obesity; Metabolic Syndrome; Hypertension (HTN); Vascular Resistance; High Blood Pressure
Keywords: Mean Arterial Pressure; Peripheral Hemodynamics; Physical Therapy; Long Term Hypertension; Resistant HTN; Systolic Blood Pressure (SBP); Diastolic Blood Pressure (DBP); Heart Rate Variability (HRV)
MeSH Terms: conditions — Essential Hypertension; Obesity, Abdominal; Metabolic Syndrome; Hypertension | interventions — Transcutaneous Electric Nerve Stimulation; Exercise; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: A randomized, two-arm, parallel-group interventional study. Participants with resistant hypertension are assigned to one of two groups. The Experimental Group receives a combined intervention consisting of Transcutaneous Electrical Stimulation (TENS) and Isometric Exercise. The Control Group receives a conventional physical therapy program. Both groups follow their respective protocols concurrently for a period of [Insert Number] weeks, with peripheral hemodynamic parameters assessed at baseline and following the completion of the intervention."
Who Masked: Outcomes Assessor
Masking Description: The study follows a single-blind design. While the participants and the physical therapist providing the treatment are aware of the group allocation due to the nature of the interventions (isometric exercise and TENS), the outcomes assessor will remain blinded. This individual, responsible for measuring peripheral hemodynamic parameters at baseline and post-intervention, will not have access to the randomization list or the participants' group assignments. Additionally, the data analyst will be blinded by using coded identifiers for the groups during statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined TENS and Isometric Exercise (Experimental): Participants in this arm will receive a combined intervention of Transcutaneous Electrical Nerve Stimulation (TENS) and a structured protocol of isometric exercises specifically designed for patients with resistant hypertension.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Behavioral: Isometric Exercise
- Conventional Physical Therapy Program (Active Comparator): Participants in this arm will receive a standard conventional physical therapy program. This serves as the active control to compare the effectiveness of the combined TENS and exercise protocol against current standard practice.
  Interventions: Behavioral: Aerobic, Dynamic Resistance, stretch and Breathing Exercises and Lifestyle Modification Advices

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — Application of TENS Electrode placements: bilaterally over the Paraspinal muscles at the T1-T5 levels (upper thoracic region), targeting sympathetic outflow to the cardiovascular system.
  Frequency: 2-10 Hz (low frequency stimulation) Pulse duration: 200 microseconds Intensity: strong but comfortable tingling sensations, below motor threshold (typically between 10-20mA) Session duration: 30 minutes per session Session frequency: 3 times per week Total intervention duration: 8 weeks
  Arms: Combined TENS and Isometric Exercise
Behavioral: Isometric Exercise — Device: Hand grip dynamometer. protocol:
  * 30% of the participants' maximal voluntary contraction (MVC).
  * Duration per trial: 2 minutes.
  * Number of trials per session: 4 repetitions
  * Rest interval between trials: 1 minute
  * Session frequency: 3 sessions per week
  * Total session duration: 14 minutes
  Per session:
  * 4 sets × 2 minutes = 8 minutes of active contraction
  * Rest between sets: 1 to 3 minutes (average 2 min × 3 rests = 6 minutes)
  * So total session time: average 14 minutes. • Total intervention duration: 8 weeks
  Arms: Combined TENS and Isometric Exercise
Behavioral: Aerobic, Dynamic Resistance, stretch and Breathing Exercises and Lifestyle Modification Advices — 1. Aerobic exercise: moderate (brisk walking): 30 min, 5 times per week.
  2. Engage in dynamic resistance exercise (weight training): 2 or more days non-consecutive.
  3. Minimize sedentary behavior
  4. Maintain healthy weight
  5. Nutritional advice like:
     * Eat at least 5 portions of fruit and vegetables
     * Eat more lean protein e.g. Fish and nuts
     * Eat less salt <5g or 1tsp
     * Eat 25-29 g of fiber
     * Limit alcohol
     * Drink 2-3 cups of coffee and/or tea (unsweetened)
  6. Others:
     * Sleep: 7-9h/day
     * Reduce stress: practice meditation or yoga 30 min per day
     * Listen to music at least 25 min, 3 times per week
     * Stop smoking
     * Limit pollutions exposure
     * Use digital wearables/apps to track movement
  7. Breathing exercise:
     Slow breathing at a rate of 6 breath/min for 10 minutes.
  8. Stretching exercise:
  Static stretching exercise is mainly for large bulky muscles 30 sec stretch, 30 sec rest for 5 min
  Arms: Conventional Physical Therapy Program

SUMMARY:
The goal of this clinical trial is to learn if the combination between transcutaneous electrical nerve stimulation (TENS) and isometric exercise (IE) can improve blood pressure in men and women between 50 to 60 years old suffered from resistant hypertension which is a type of hypertension where blood pressure remains above your target goal despite the use of three or more different classes of antihypertensive medications at their maximum tolerated doses. The main question to answer is:

Is there a significant effect on the combined use of TENS and IE on peripheral hemodynamic parameters in patients with resistant hypertension? Total sample will be 50 patients from both sexes

I will compare between two groups:

Experimental group (15 men, 10 women) will take: medication plus IE and TENS Control group (15 men, 10 women) will take: medication plus Conventional Physical Therapy Program

DETAILED DESCRIPTION:
1. Study Rationale: Resistant hypertension (RH) remains a significant clinical challenge, often requiring four or more medications to achieve blood pressure control. Chronic sympathetic overactivity is a hallmark of RH. (TENS) has shown promise in modulating autonomic tone, while IE is known to improve endothelial function and vascular resistance. However, the combined effect of these two non-pharmacological interventions on peripheral hemodynamics in RH patients has not been fully explored.
2. Objectives: The primary objective of this study is to investigate the effect of a combined program of TENS and IE on peripheral hemodynamic parameters, including (Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Pressure (MAP), Pulse Pressure (PP) and Heart Rate Variability (HRV) in patients diagnosed with RH.
3. Study Design and Procedures: 50 Participants from both sexes will be randomly assigned using closed envelop to either the Experimental Group (Combined Intervention) or the Control Group (Conventional physical therapy program)

<!-- -->

1. Experimental group TENS protocol It will be used to stimulate the cervicothoracic sympathetic outflow (C7-T4), which contributes to the modulation of sympathetic activity, a key factor in the pathophysiology and management of resistant hypertension (RH) Electrode placements: bilaterally over the Paraspinal muscles at the T1-T5 levels (upper thoracic region), targeting sympathetic outflow to the cardiovascular system.

   -Frequency: 2-10 Hz (low frequency stimulation)

   -Pulse duration: 200 microseconds

   -Intensity: strong but comfortable tingling sensations, below motor threshold (typically between 10-20mA)

   -Session duration: 30 minutes per session

   -Session frequency: 3 times per week

   -Total intervention duration: 8 weeks IE protocol Handgrip Dynamometer: It will be used for isometric exercise training. The majority of IET research has utilized a handgrip (dynamometer) protocol, generally performed at 30% of the participant's maximal voluntary contraction (MVC)

   -Hand grip dynamometer.

   -30% of the participants' maximal voluntary contraction (MVC).

   -Duration per trial: 2 minutes.

   -Number of trials per session: 4 repetitions

   -Rest interval between trials: 1 minute

   -Session frequency: 3 sessions per week

   -Total session duration: 14 minutes
2. Control group Conventional physical therapy programs

   * Aerobic exercise The control group will participate in a supervised overground brisk walking program, which serves as the contemporary standard of care for non-pharmacological blood pressure management. The program is designed to meet the latest physical activity clinical practice guidelines for hypertensive populations.

   Setting and Monitoring sessions will be conducted in a climate-controlled, flat-surface indoor corridor. To ensure the accuracy of the prescribed intensity, participants will be equipped with a digital heart rate monitor (pulse oximeter) and a stopwatch. Baseline hemodynamic parameters, including resting blood pressure and heart rate, will be recorded before each session to ensure patient stability.

   Brisk Walking Protocol The intervention will be performed three times per week for eight consecutive weeks. Each session is structured into three distinct phases (Lopes et al., 2021).

   Warm-up Phase (5 minutes): Participants will engage in low-intensity walking at a self-selected pace, integrated with dynamic mobilization exercises for the lower limbs to enhance neuromuscular readiness.

   Conditioning Phase (20-30 minutes): Participants will perform brisk walking at moderate intensity. This intensity is defined as 50% to 70% of the age-predicted maximum heart rate (220 - age). According to recent consensus, this level of exertion corresponds to a score of 11 to 13 on the Borg Rating of Perceived Exertion (RPE) scale.

   Cool-down Phase (5 minutes): The session will conclude with gradual deceleration and static stretching of the major muscle groups (quadriceps, hamstrings, and gastrocnemius) to facilitate the gradual return of heart rate to baseline and prevent post-exercise syncope.

   - Dynamic resistance exercise (weight training): Patients in the control group will undergo a standardized, supervised Dynamic Resistance Training (DRT) program. This protocol is designed based on the AHA/ACSM guidelines for hypertensive patients, focusing on large muscle groups with minimal equipment to ensure safety and clinical reproducibility.

1. Exercise Parameters (FITT Principle) Frequency: 3 sessions per week on non-consecutive days. Intensity: Moderate intensity, defined as 40%-50% of 1-Repetition Maximum (1-RM) or a Rating of Perceived Exertion (RPE) of 11-13 on the Borg Scale (Fairly Light to Somewhat Hard).

Time: Approximately 30-40 minutes per session. 2. Exercise Selection

The circuit consists of simple, functional movements to improve peripheral vascular conductance:

Lower Body: Partial Squats (using a chair for support) and Calf Raises. Upper Body: Dumbbell Chest Press (supine) and Bicep Curls. Core: Pelvic Tilts (supine) to avoid intra-abdominal pressure spikes. 3. Structure of the Session Warm-up: 5 minutes of low-intensity walking or active range of motion exercises.

Conditioning Phase: 2-3 sets of 10-12 repetitions for each exercise. Rest Periods: A mandatory 90-second rest between sets to prevent cumulative blood pressure elevation.

Breathing Technique: Patients are strictly instructed to use rhythmic breathing (exhale during exertion) to avoid the Valsalva maneuver.

Cool-down: 5 minutes of static stretching and deep breathing exercises. -Stretching exercise A standardized static stretching program will be implemented. This protocol follows the ACSM guidelines to improve the range of motion and facilitate a reduction in systemic vascular resistance.

1. Stretching Parameters Type: Static stretching (passive and active-assisted). Frequency: 3 days per week (integrated at the end of each exercise session). Intensity: Stretch to the point of "mild discomfort" or "feeling of tightness," but not pain.

Duration: Each stretch is held for 30 seconds. Volume: 2 repetitions for each muscle group. 2. Muscle Groups Targeted

The focus is on large muscle groups to maximize the effect on peripheral blood flow:

Lower Body:

Hamstrings: Seated toe touch or supine hamstring stretch. Gastrocnemius (Calf): Wall-supported calf stretch. Quadriceps: Standing or side-lying quad stretch.

Upper Body:

Pectoralis: Doorway chest stretch (to improve thoracic expansion). Upper Trapezius: Gentle neck lateral flexion. Triceps: Overhead triceps stretch. - Breathing Exercise This protocol is designed to be performed at the beginning or end of each session to promote systemic vasodilation.

1. Technique: Diaphragmatic Breathing (Paced Breathing) Position: Patients are placed in a comfortable supine position with knees slightly bent or seated in a supportive chair.

   Procedure:

   The patient places one hand on the upper chest and the other on the abdomen (just below the rib cage).

   Inhalation: Breathe slowly through the nose for 4 seconds, ensuring the abdomen rises while the chest remains relatively still.

   Exhalation: Breathe out slowly through pursed lips for 6 seconds. Breathing Rate: Aim for 6 breaths per minute (this frequency is specifically shown to optimize baroreflex sensitivity).
2. Parameters Frequency: 3 sessions per week (integrated into the physical therapy program). Duration: 10-15 minutes per session. Intensity: Effortless and relaxed; the patient should not feel short of breath or strained.
3. Clinical Monitoring The physical therapist monitors the patient for any signs of dizziness or hyperventilation.

Emphasis is placed on the prolonged exhalation phase, which triggers the relaxation response and reduces peripheral vascular resistance.

-General Advice for Both Groups: Minimize sedentary behavior Maintain a healthy weight

Nutritional advice like:

Eat at least 5 portions of fruit and vegetables Eat more lean protein e.g. Fish and nuts Eat less salt <5g or 1tsp Eat 25-29 g of fiber Limit alcohol Drink 2-3 cups of coffee and/or tea (unsweetened)

Others:

Sleep: 7-9h/day Reduce stress: practice meditation or yoga 30 min per day Listen to music at least 25 min, 3 times per week Stop smoking Limit pollutions exposure Use digital wearables/apps to track movement

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 60 years. Both sexes were included Patients had been diagnosed with hypertension for at least 5 years.

Patients had resistant hypertension according to (Whelton et al 2018), defined as:

* Systolic blood pressure (SBP) ≥140 mmHg and/or diastolic blood pressure (DBP) ≥90 mmHg despite the use of three or more antihypertensive medications of different classes, including a diuretic,
* or controlled blood pressure (<140/90 mmHg) while on four or more antihypertensive medications.

Body Mass Index (BMI) 25: 34.9 kg/m²

Increased waist circumference, defined as:

* Greater than 102 cm for males.
* Greater than 88 cm for females.

Exclusion Criteria:

* Secondary hypertension due to identifiable causes (e.g., renal artery stenosis, primary aldosteronism, pheochromocytoma).
* History of major cardiovascular events in the last 6 months (e.g., myocardial infarction, stroke, or heart failure exacerbation).
* Severe musculoskeletal or neurological disorders that impair the ability to perform isometric exercise safely (e.g., recent joint replacement, severe osteoarthritis, stroke with residual motor deficit).
* Contraindications to the use of Transcutaneous Electrical Nerve Stimulation (TENS):

Implanted electronic devices: pacemakers, cardioverter defibrillators. Uncontrolled arrhythmias. Sever skin condition: open wounds, rashes, burns, eczema. Peripheral neuropathy or sensory loss.

-Known cognitive impairment or psychiatric conditions that would limit the ability to follow instructions or provide informed consent.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Pulse Pressure | 8 weeks
  Definition and Calculation: Pulse Pressure (PP) is the primary hemodynamic outcome, representing the pulsatile component of the blood pressure waveform. It is calculated as the difference between Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP): PP = SBP - DBP.
  Measurement Method: Measurements will be obtained via manual auscultation using a calibrated sphygmomanometer. SBP is identified at Korotkoff Phase I and DBP at Phase V. To ensure precision, three readings will be taken at 2-minute intervals after a 5-minute rest; the mean values will be used for the final PP calculation.
  Clinical Significance: In resistant hypertension, PP is a robust indicator of large-artery stiffness and cardiovascular risk. This study evaluates the effect of combined transcutaneous electrical stimulation and isometric exercise on reducing PP, signifying improved vascular compliance and reduced hemodynamic load.
  Unit of Measure: mmHg
Mean Arterial Blood Pressure | 8 weeks
  Description: The primary outcome is the change in Mean Arterial Pressure (MAP) from baseline to the end of the intervention. MAP represents the average arterial pressure during a cardiac cycle, serving as a critical indicator of hemodynamic load in patients with resistant hypertension.
  Measurement & Calculation: MAP will be determined via the manual auscultatory method using a mercury and a stethoscope.
  Following a 10-minute quiet rest in a seated position, three readings will be taken from the non-dominant arm (2-minute intervals).
  SBP and DBP will be recorded at Korotkoff phases I and V. MAP will then be calculated using the formula: MAP = DBP + 1/3(SBP - DBP).
  Unit of Measure: mmHg
Systolic Blood Pressure (SBP) | 8 weeks
  Definition: Systolic Blood Pressure (SBP) is the primary measure of peripheral hemodynamics. SBP reflects the maximum pressure exerted against arterial walls during ventricular contraction, while DBP reflects the minimum pressure during ventricular relaxation.
  Measurement Protocol: Measurements will be performed via manual auscultation using a calibrated sphygmomanometer and a high-quality stethoscope. SBP will be recorded at the onset of Korotkoff Phase I (clear tapping). Participants will rest seated for 5 minutes prior to assessment. Three readings, separated by 2-minute intervals, will be averaged to determine the final values.
  Clinical Significance: In resistant hypertension, SBP is the gold-standard markers for evaluating the efficacy of the combined transcutaneous electrical stimulation and isometric exercise intervention in reducing systemic vascular resistance and cardiovascular load.
  Unit of Measurement: mmHg
Heart Rate | 8 weeks
  Definition: Heart Rate (HR), measured in beats per minute (BPM), serves as a primary indicator of autonomic nervous system activity and cardiovascular workload. In patients with resistant hypertension, it reflects the chronotropic response to the combined intervention.
  Measurement Method: HR will be measured using a Granzia Pulsox digital pulse oximeter.
  The device will be placed on the index finger of the participant's non-dominant hand. Following a 5-minute period of seated rest, the investigator will wait for a stable plethysmographic signal on the Granzia display before recording the value. To ensure reliability, three consecutive readings will be taken at 1-minute intervals, and the mean value will be used as the primary data point for analysis.
  Clinical Significance: A reduction in resting HR would indicate a successful modulation of sympathetic activity following the TENS and isometric exercise protocol.
Diastolic Blood Pressure (DBP) | 8 weeks
  It is the primary measure of peripheral hemodynamics. DBP reflects the minimum pressure during ventricular relaxation.
  Measurement Protocol: Measurements will be performed via manual auscultation using a calibrated sphygmomanometer and a high-quality stethoscope. DBP will be recorded at the onset of Korotkoff at Phase V (disappearance of sound). Participants will rest seated for 5 minutes prior to assessment. Three readings, separated by 2-minute intervals, will be averaged to determine the final values.
  Clinical Significance: In resistant hypertension, DBP is the gold-standard markers for evaluating the efficacy of the combined transcutaneous electrical stimulation and isometric exercise intervention in reducing systemic vascular resistance and cardiovascular load.
  Unit of Measurement: mmHg

SECONDARY OUTCOMES:
Autonomic parameters: Heart Rate Variability | 8 weeks
  Definition: Heart Rate Variability (HRV) is the physiological variation in time intervals between consecutive heartbeats (RR intervals). It is a non-invasive marker of autonomic regulation; high HRV indicates parasympathetic dominance (relaxation), while low HRV is associated with sympathetic overactivity and increased cardiovascular risk in hypertensive patients.
  Measurement Method: HRV will be assessed using the Welltory application via smartphone photoplethysmography (PPG). Participants will place their index finger over the phone's camera and flash for a 2-minute "liquid" measurement. To ensure clinical-grade data, the app's 300-beat mode will be enabled to capture time-domain (e.g., SDNN, RMSSD) and frequency-domain (LF/HF ratio) metrics.
  Standardization: Measurements will be performed at baseline and post-intervention in a seated, quiet environment. The mean of two consecutive measurements with >95% accuracy scores (as reported by Welltory) will be used for analysis.
Physiological parameters: Oxygen Saturation | 8 weeks
  Definition: Peripheral oxygen saturation ($SpO_2$) measures the percentage of oxygen-saturated hemoglobin. In this trial, it serves as a safety and physiological marker during the combined TENS and isometric exercise intervention for resistant hypertension.
  Measurement Method: SpO_2 will be measured using a Granzia digital pulse oximeter. The sensor will be applied to the index finger of the non-dominant hand. Following 5 minutes of seated rest, the investigator will record the value once a stable plethysmographic waveform is displayed on the Granzia screen. Three readings will be averaged to ensure data reliability.
  Clinical Significance: Monitoring SpO_2 ensures that the pressor response during exercise does not compromise systemic oxygenation. Normal values (> 95) indicate the intervention is well-tolerated without respiratory distress.
Functional parameter: QoL (SF-36) | 8 weeks
  Description: The Short Form-36 (SF-36) questionnaire is used to evaluate the physical and mental health status. It consists of 36 items covering eight health domains.
  Unit of Measure: Units on a scale Scale Range: The total score ranges from 0 to 100. Interpretation: Higher scores indicate better health-related quality of life, while lower scores indicate more disability or poorer health status.
Functional Capacity (modified Harvard step test) | 8 weeks
  Description: The Modified Harvard Step Test is used to measure cardiovascular fitness and aerobic capacity. The Fitness Index is calculated based on the duration of the test and the heart rate recovery after exercise.
  Unit of Measure: Units on a scale Scale Range: Fitness Index scores (typically range from <55 "Poor" to >90 "Excellent").
  Interpretation: A higher Fitness Index score reflects better cardiovascular endurance and more

CONTACTS AND LOCATIONS:
Locations (1):
- Out Clinics of Port Said Hospitals, Port Said, Port Said Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No